CLINICAL TRIAL: NCT07283016
Title: Effects of Pectoralis Minor Stretching and Strengthening Exercises on Shoulder Pain, Scapular Dyskinesis and Thoracic Expansion Among Patients With Adhesive Capsulitis: A Randomized Controlled Trial
Brief Title: Effects of Pectoralis Minor Exercises on Shoulder Pain, Scapular Dyskinesis and Thoracic Expansion in Adhesive Capsulitis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/030
Record Dates: First submitted 2025-11-24; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Adhesive Capsulitis
Keywords: Strengthening exercises; Scapular dyskinesis; Shoulder Pain; Thoracic Expansion; Pectoralis minor
MeSH Terms: conditions — Bursitis; Shoulder Pain | interventions — Range of Motion, Articular

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Pectoralis Minor Stretching and Strengthening with Mobility and Stability Exercises
  Interventions: Other: Pectoralis Minor Stretching and Strengthening with Mobility and Stability exercises
- Control group (Active Comparator): Mobility and Stability Exercises
  Interventions: Other: Mobility and Stability exercises

INTERVENTIONS:
Other: Pectoralis Minor Stretching and Strengthening with Mobility and Stability exercises — Participants in this group will follow a 6 week program targeting the Pectoralis Minor exercises in addition to mobility and stability exercises as explained in the control group used for adhesive capsulitis management. Pectoralis minor exercises include pectoralis minor stretching and strengthening. Pectoralis minor stretching exercises are unilateral corner and foam roller stretches (4 repetitions × 30 seconds hold, with a 30-second rest, performed 4 days a week for 6 weeks) to improve chest mobility. Pectoralis minor strengthening exercises are scapular push-ups (protraction-focused), scapular protraction with resistance bands, and wall slides with scapular protraction (3 sets × 10 repetitions, performed 4 days a week for 6 weeks) to boost muscle strength and support proper scapular movement. These interventions aim to reduce shoulder pain, improve scapular function, and enhance chest compliance in patients with adhesive capsulitis.
  Arms: Experimental Group
Other: Mobility and Stability exercises — Participants in the control group will receive a standardized physical therapy protocol commonly used for adhesive capsulitis management over a period of 6 weeks. This will include mobility and stability exercises. Mobility Exercises are passive range-of-motion exercises combined with joint mobilization techniques such as pendulum exercises, wall crawls, and towel stretches (3 sets of 10 repetitions of each exercise, performed 4 days a week for 6 weeks). Stability Exercises are isometric rotator cuff exercises performed (3 sets of 10 repetitions of each exercise, performed 4 days a week for 6 weeks). This basic treatment approach aims to reduce pain, improve joint mobility, and support gradual recovery in adhesive capsulitis without specifically targeting the pectoralis minor.
  Arms: Control group

SUMMARY:
The goal of the current study is to evaluate the effects of pectoralis minor stretching and strengthening with mobility and stability exercises in patients aged 40-70 years with adhesive capsulitis. The main questions it aims to answer are:

Does the combination of pectoralis minor stretching and strengthening with mobility and stability exercises significantly reduce shoulder pain compared to mobility and stability exercises only? Does the combination of pectoralis minor stretching and strengthening with mobility and stability exercises improve scapular dyskinesis (scapular movement patterns) and thoracic expansion more effectively than mobility and stability exercises? Participants will be assigned to either an experimental group receiving pectoralis minor stretching and strengthening exercises with mobility and stability exercises or a control group receiving mobility and stability exercises only, and will complete standardized assessments of shoulder pain, scapular dyskinesis (scapular movement patterns) and thoracic expansion before and after the intervention.

DETAILED DESCRIPTION:
This clinical trial is designed to evaluate the combined effects of pectoralis minor stretching and strengthening with mobility and stability exercises on shoulder pain, scapular dyskinesis (scapular movement patterns) and thoracic expansion in individuals with adhesive capsulitis. It is commonly linked to reduce pectoralis minor tightness and improve pectoralis minor strength and interventions that target both mobility and stability as well as pectoralis minor correction may offer improved clinical outcomes of shoulder pain, scapular dyskinesis (scapular movement patterns) and thoracic expansion. All participants will undergo baseline assessment, including shoulder pain measured with the Numeric Pain Rating Scale, scapular dyskinesis assessed using the modified scapular assistance test, and thoracic expansion measured using a cloth measuring tape.

Participants will be randomized into two groups (Control Group and Experimental Group). Participants in the control group will perform mobility and stability exercises. Mobility Exercises are passive range-of-motion exercises combined with joint mobilization techniques such as pendulum exercises, wall crawls, and towel stretches. Stability Exercises are isometric rotator cuff exercises. Participants in the experimental group will perform mobility and stability exercises as described in the control group, plus pectoralis minor exercises. Pectoralis minor stretching exercises are unilateral corner and foam roller stretches. Pectoralis minor strengthening exercises are scapular push-ups (protraction-focused), scapular protraction with resistance bands, and wall slides with scapular protraction.

The interventions will occur 4 times per week for 6 weeks, with each session lasting approximately 30-40 minutes. Participants will be advised to avoid any external treatments during the study period. Post-intervention assessments will be conducted immediately after six weeks post intervention. This study aims to clarify whether the integration of pectoralis minor exercises results in superior clinical outcomes compared to mobility and stability exercises alone in the management of adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 - 70 years
* Gender: Both Male & Female
* Clinical diagnosis of adhesive capsulitis (Thawing stage).
* Reduced thoracic expansion.
* Scapular dyskinesis

Exclusion Criteria:

* Presence of rotator cuff tear, labral tears, or glenohumeral arthritis confirmed through imaging
* Post-stroke hemiparesis,
* Winged scapula due to lesions of long thoracic nerve or spinal accessory nerve.
* Rotator cuff repair
* Capsular release
* Arthroplasty

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain | From enrollment to the end of treatment at 6 weeks
  Shoulder pain intensity is assessed using the Numeric Pain Rating Scale. The Numeric Pain Rating Scale functions as a basic method to examine pain severity. It is a unidimensional measure where participants rate their pain on an 11-point scale. The scale ranges from 0 to 10, where 0 represents "no pain" and 10 represents "worst pain imaginable". The assessment tool is available through spoken language or visual presentation, enabling smooth clinical application. Participants select the number that best represents their current level of discomfort, with higher scores indicating greater levels of pain intensity.

SECONDARY OUTCOMES:
Scapular Dyskinesis | From enrollment to the end of treatment at 6
  Scapular dyskinesis is evaluated using the Modified Scapular Assistance Test. The Modified Scapular Assistance Test functions as a clinical evaluation method for determining how scapular dyskinesis affects shoulder pain symptoms. During the test, the examiner provides manual assistance to both upward scapular rotation and scapular posterior tilting as the patient performs shoulder arm elevation. The test result is determined by the change in pain symptoms. The test becomes positive when the pain decreases by two points or more during motion assistance compared to unassisted movement, pointing to scapular motion dysfunction as a potential symptomatic factor.
  The Modified Scapular Assistance Test is not a numerical scoring test. It is a qualitative value. It is positive when the patient's shoulder pain decreases and it is negative when the shoulder Pain does not decrease.
Thoracic expansion | From enrollment to the end of treatment at 6
  Thoracic expansion is measured using a cloth measuring tape. This serves as a practical clinical method to assess chest wall movement and respiratory function. Measurements are taken at three specific anatomical levels: the axilla, the fourth intercostal space, and the xiphoid level. The difference in chest circumference between full expiration and full inspiration is recorded for each level. Higher values representing the difference between inspiration and expiration indicate greater thoracic mobility and chest expansion.

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD TARIQ RAFIQ, Principal Investigator — Lahore University of Biological & Applied Sciences

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared after completion of the study
Supporting Information: Study Protocol, CSR
Time Frame: After completion of the study until the time of 5 years.